CLINICAL TRIAL: NCT03203798
Title: Effects of Pelvic Floor Muscle Training or Hipopressive Abdominal Gymnastics in the Treatment of Women's Stress Urinary Incontinence: a Prospective, Randomized, Controlled Study
Brief Title: Effects of Training of Pelvic Floor Muscles (MAP) on Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Luciene Aparecida José Vaz, Principal Investigator, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.516.103
Record Dates: First submitted 2017-06-26; First posted 2017-06-29 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training of pelvic floor muscles (Active Comparator)
  Interventions: Procedure: Training of pelvic floor muscles
- Hipopressive abdominal gymnastics (Experimental)
  Interventions: Procedure: Hipopressive abdominal gymnastics

INTERVENTIONS:
Procedure: Training of pelvic floor muscles — The pelvic floor muscle training group will be composed of randomized women and participated for 12 weeks of intervention, where it was performed in groups of a maximum of 4 patients, starting in the first 4 weeks with 3 sets of 8 repetitions of contraction maintained for 5 seconds In antigravity postures, with two lying postures and one sitting posture, and evolving to the next 4 weeks for 3 sets with 10 repetitions of contraction maintained for 5 seconds being a lying posture, a seated posture and orthostatic posture in the last 4 weeks 3 Series of 12 repetitions of contraction maintained for 5 seconds in the gravitational postures, being one sitting posture and two orthostatic postures.
  Arms: Training of pelvic floor muscles
Procedure: Hipopressive abdominal gymnastics — The hipopressiva abdominal gymnastics group will be composed of randomized women who participated for 12 weeks of intervention, where it was performed in groups of a maximum of 4 patients, being performed respecting the basic sequence of the exercise proposed by Marcel Caufriez: 1) Inspiration, 2) Maximum Expiration, 3) Diaphragmatic aspiration being performed 3 series of 8 to 12 repetitions. The exercises will be performed in groups of a maximum of 4 patients, starting in the first 4 weeks with 3 sets of 8 repetitions in antigravity postures, with two lying postures and one sitting posture, and evolving over the next 4 weeks to 3 sets with 10 repetitions A lying posture, a sitting posture and orthostatic posture, in the last 4 weeks 3 sets of 12 repetitions in the gravitational postures, being a sitting posture and two orthostatic postures.
  Arms: Hipopressive abdominal gymnastics

SUMMARY:
In the current scientific literature, it is clear that SUI can cause several social, hygienic and personal relationship problems. It has also been proven that this condition affects many more menopausal women than menacme, and this is believed to be due to the hypoestrogenism characteristic of this phase.

On the other hand, weakness of the pelvic floor muscles (PFM) is also related to the genesis of SUI. The role of these muscles would be to keep the bladder neck elevated (above the pubic symphysis) during increases in abdominal pressure, and its weakness would lead to excessive lowering of the bladder neck at these times, leading to SUI due to bladder neck hypermobility.

The conservative treatment of this condition, therefore, encompasses the strengthening of PFMs, which would avoid excessive descent of the bladder neck during increases in abdominal pressure, thereby reducing urinary loss.

In the current literature there are studies proving the effectiveness of pelvic floor muscle training; however, in relation to the literature on abdominal hipopressive gymnastics, it is observed that the scientific evidence is still poor, however, the technique is still Widely spread through extension courses offered throughout Latin America, France and Spain; With regard to the comparison of these methods with respect to their clinical efficacy and the quality of life and patient satisfaction, there are no consistent studies, and this fact motivated us to carry out this study.

ELIGIBILITY:
Inclusion Criteria:

* Women with IUE and with a modified Oxford scale of at least 1.

Exclusion Criteria:

* Presence of neuromuscular diseases
* Uncontrolled diabetes

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-09-26 (Actual); Study Completion 2020-08-26 (Estimated)

PRIMARY OUTCOMES:
Check for modification on modified oxford scale | two months
  Bidigital palpation will be performed in the vagina and requested the maximum voluntary contraction of the pelvic floor muscles.
Check for modification on Perineometry | two months
  A silicone probe will be introduced into the vaginal cavity, and then it will be inflated to 100 cm / H2O, and reset. After this will be requested the maximum voluntary contraction maintained for 5 seconds, with interval of 1 minute to rest and after it will be repeated twice.

SECONDARY OUTCOMES:
International Consultation on Incontinence Questionnaire Short Form | two months
  Self-administered questionnaire to evaluate the impact of incontinence on the life of the research participant.
Pelvic Floor Impact Questionnaire (PFIQ-7) Floor Impact Questionnaire (PFIQ-7) | two months
  A self-administered questionnaire that presents seven questions to evaluate the impact of each subsession on the participant's quality of life.
Pelvic Floor Distress Inventory (PFDI-20) | two months
  A self-administered questionnaire composed of 20 questions applied to assess the impact of each domain on the life of the research participant.
Void diary | two months
  Diary delivered to the participant to note for seven days the urinary frequency daytime, night, amount of loss and exchange of absorbents if you use.

CONTACTS AND LOCATIONS:
Overall Officials: Luciene Aparecida Vaz, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Luciene Aparecida José Vaz, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322